CLINICAL TRIAL: NCT03357848
Title: Impact of Caloric and Protein Adequacy on Postoperative Clinical Outcomes of Patients Undergoing Major Abdominal Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, Professor/ Nutrition Service Coordinator, Federal University of Minas Gerais
Other Study IDs: CAAE-12279713.1.0000.5149
Record Dates: First submitted 2017-11-22; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Surgery; Postoperative Complications; Cancer; Energy Supply; Deficiency
MeSH Terms: conditions — Postoperative Complications; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Surgical patients receiving nutritional support (enteral and/or parenteral nutrition) pre and/or after surgery
- Control group: Surgical patients without nutritional support during the perioperative period

SUMMARY:
The role of nutritional therapy (TN) in the surgical patient is well described in the literature and is associated with reductions in postoperative complications, length of hospital stay, and mortality. Adequate determination of caloric and protein requirements is an essential step in the TN institution, avoiding hypoalimentation and hyperalimentation. Thus, it is essential to understand the changes in energy expenditure after surgery and its relation with nutritional status. In addition, little is known about the effect of nutritional therapy and caloric adequacy on parameters such as phase angle and dynamometry. Thus, the objective of this study is to evaluate the changes in energy expenditure after major abdominal surgeries and to evaluate the phase angle and dynamometry as possible markers of nutritional therapy. Energy expenditure will be assessed by indirect calorimetry. Functionality will be assessed by means of dynamometry and 6-minute walk test. Nutritional diagnosis will be given through subjective global assessment. Energy and protein intake will be monitored and registered daily. Phase angle will be obtained by performing bioelectrical impedance.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Patients admitted for major abdominal surgery
* Sign the consent form

Exclusion Criteria:

* Length of hospital stay less than 3 days
* Pregnancy
* Patients who, for any reason, can not perform indirect calorimetry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major abdominal surgery at the University Hospital of University Federal of Minas Gerais
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-12-19 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 30 days after surgery
  According to the Dindo-Clavien protocol

SECONDARY OUTCOMES:
Phase angle | 24 hours pre-surgery, 3 and 7 days after surgery
  Changes in phase angle after surgery as measured by bioelectrical impedance
Body composition | 24 hours pre-surgery, 3 and 7 days after surgery
  Changes in body composition after surgery as measured by bioelectrical impedance
Nutritional status | 24 hours pre-surgery and 7 days after surgery
  Changes in nutritional status after surgery as assessed by subjective global assessment (SGA)
Functional status | 24 hours pre-surgery, 3 and 7 days after surgery
  Changes in functional status after surgery as assessed by hand grip strength
Energy expenditure | 3, 5 and 7 days after surgery
  Changes in energy expenditure after surgery measured by indirect calorimetry

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Clinics of the University Federal of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil